CLINICAL TRIAL: NCT00994708
Title: The Effect of Esomeprazole and Nissen Fundoplication on Bronchial Responsiveness, Quality of Life, Exhaled Nitric Oxide and Pulmonary Function in Patients With Gastroesophageal Reflux Disease
Brief Title: The Effect of Esomeprazole and Fundoplication on Airways
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Tampere University Hospital (Other)
Other Study IDs: R04002M
Record Dates: First submitted 2009-10-12; First posted 2009-10-14 (Estimated); Last update posted 2009-10-14 (Estimated); Status verified 2009-10

CONDITIONS: Airway Responsiveness
MeSH Terms: interventions — Esomeprazole

INTERVENTIONS:
Drug: esomeprazole

SUMMARY:
Evaluate the prevalence of bronchial responsiveness (BHR) among patients with gastroesophageal reflux disease (GERD).

Investigate correlation between bronchial reactivity and the severity of GERD, and similarly investigate the correlation between exhaled nitric oxide (NO) and the severity of GERD.

Compare the effects of esomeprazole 40 mg twice daily and Nissen fundoplication on bronchial reactivity, exhaled NO, pulmonary function and quality of life.

ELIGIBILITY:
Inclusion Criteria:

1. Over 18 of age
2. Diagnosis of gastroesophageal reflux disease
3. Compliance to perform methacholine inhalation challenge (judged by the investigator)

Exclusion Criteria:

1. Known allergy to esomeprazole or any other PPI
2. Use of systemic corticosteroids within 3 weeks before any study visit
3. Pregnancy (in a written informed consent patients are asked to assure that they are not pregnant and they are also told to immediately stop the study medication if they become pregnant during the study)
4. Incapability to keep a 3-week washout with usual antireflux medication prior to the first visit
5. Regular use of PPI or H2-RA medication 3 months after fundoplication

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 2004-12

CONTACTS AND LOCATIONS:
Locations (1):
- Tampere University Hospital, Tampere, Pirkanmaa, Finland

REFERENCES:
- [Derived] Kiljander T, Rantanen T, Kellokumpu I, Koobi T, Lammi L, Nieminen M, Poussa T, Ranta A, Saarelainen S, Salminen P. Comparison of the effects of esomeprazole and fundoplication on airway responsiveness in patients with gastro-oesophageal reflux disease. Clin Respir J. 2013 Jul;7(3):281-7. doi: 10.1111/crj.12005. Epub 2012 Oct 24. PMID 23006321